CLINICAL TRIAL: NCT04056559
Title: Normative Assessment of Adaptable Mouthguards.
Acronym: ENORMPIBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CHU Bx 2011/04
Record Dates: First submitted 2019-08-13; First posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Oral Manifestations
Keywords: Prototype; Adaptable mouthguards
MeSH Terms: conditions — Oral Manifestations

STUDY DESIGN:
Intervention Model Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIngle arm (Experimental): The research is based on a population of men and women practicing a sport at risk of oral trauma.
  Interventions: Device: Adaptable mouthguards

INTERVENTIONS:
Device: Adaptable mouthguards — Validate a prototype of Adaptable Intra-Oral Protections patented by Bordeaux University and Bordeaux University Hospital according to 3 levels (ventilation, comfort, cervical muscle activity).

SUMMARY:
The aim of this study is to the validate adaptable mouthguards prototypes, patented by Bordeaux University and Bordeaux University Hospital.

DETAILED DESCRIPTION:
The current state of knowledge in the areas of mouthguards shows that type II (adaptable) models account for 90% of the mouthguards of the sporting population. But a majority of these devices do not appear to comply with the European Directive 89/686 / European Economic Community.

A previous work consisted of the production of prototypes of mouthguards meeting the essential requirements of the directive. These prototypes were the subject of a patent filed by the Bordeaux University and the Bordeaux University Hospital.

The aim of this study is to the validate the prototypes for a future launch on the market.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged 18 to 35,
* Subject affiliated to a social security,
* Subject who has signed the free and informed consent form.

Exclusion Criteria:

* Subject with a pathology incompatible with the performance of the test, namely: Recent infarction,Threat syndrome, blood pressure resting> 200/120 mmHg, uncompensated cardiac insufficiency, atrioventricular block 3rd degree acquired, Myocarditis, Pericarditis, Endocarditis, Aortic Dissection, Intracardiac Tumor or Thrombus, Deep Vein Thrombosis, Pulmonary Embolism,
* Subject under B-mimetic drug treatment,
* Subject under safeguard of justice,
* Subject participating in another search,
* Subject during pregnancy.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-09-09 (Actual); Primary Completion 2012-06-29 (Actual); Study Completion 2012-06-29 (Actual)

PRIMARY OUTCOMES:
Impact on ventilatory flow rate by minute | At Week 51
  Average of measured values in one minute, compared to maximum aerobic reference speed of the subject
  Modification of the ventilatory flow rate by min
Impact on O2 consumption | At Week 51
  Average of measured values in one minute, compared to reference of the subject
Impact on respiratory rate | At Week 51
  Average of measured values in one minute, compared to reference of the subject
Impact on current volume | At Week 51
  Average of measured values in one minute, compared to reference of the subject
Impact on CO2 production | At Week 51
  Average of measured values in one minute, compared to reference of the subject
Impact on comfort according an analogical visual scale for 11 criteria | At Week 51
  According an analogical visual scale (from 0 to 10) for 11 criteria (retention, muco-gingival appearance, mouth opening height, volume of mouthguards, nausea, phonation, open mouth ventilation, tight jaw ventilation, salivation, masticatory muscles, temporomandibular joint)
Impact on electromyographic recording | At Week 52
  The electromyographic activity will be amplified and filtered (bandwidth 10-1000 Hz). The signals will be digitized using a CED 1401 interface coupled to a microcomputer that is controlled by the "SPIKE2" software. The digitization frequency will be 2,000 Hz. The software "SPIKE2" will then calculate what is called "integrated electromyogram": the electromyographic signals will be rectified and filtered with a moving average having a period of 0,2 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe POISSON, Dr, Principal Investigator — University Hospital, Bordeaux

IPD SHARING:
Plan to Share IPD: No